CLINICAL TRIAL: NCT00309322
Title: A Phase 2, Multicenter, Randomized, Blinded, Controlled Study of NV-101 for Safety and Efficacy in Pediatric Dental Patients Undergoing Mandibular and Maxillary Procedures
Brief Title: Study of NV-101 for Safety and Efficacy in Pediatric Dental Patients Undergoing Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novalar Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NOVA 05-PEDS
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Anesthesia, Dental
Keywords: Soft Tissue Anesthesia (Numbness)
MeSH Terms: conditions — Hypesthesia | interventions — Phentolamine

INTERVENTIONS:
Drug: Phentolamine Mesylate (NV-101)

SUMMARY:
This Phase 2 clinical study is designed as a multicenter, randomized, blinded, controlled study to evaluate the safety and efficacy of NV-101 in approximately 150 children 4 to 11 years of age. NV-101 or sham injection is administered at the completion of a dental procedure requiring local anesthesia with 2% lidocaine with 1:100,000 epinephrine. The dental procedure(s) shall be performed in a single quadrant of the mouth and include cavity preparation, restoration/filling, teeth cleaning (non-surgical scaling and/or root planing), or crowns.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 4 to 11 years of age
* Sufficiently healthy, as determined by the Investigator, to receive routine dental care
* Requires a restorative procedure such as cavity preparation, or such as teeth cleaning (non-surgical scaling and/or root planing) in a single quadrant of the mouth
* Requires local anesthesia with 2% lidocaine with 1:100,000 epinephrine administered by submucosal injection
* Dental procedure(s) completed with 60 minutes of injection of local anesthetic
* Can be trained to complete the Wong Baker Pain Rating Scale
* For subjects 6 to 11 years of age who are trainable in standardized palpation procedure:

  * have normal lip sensation at baseline prior to administration of local anesthetic
  * have numbness of the relevant lip quadrant at completion of the dental procedure
* Negative urine pregnancy test at screening in female subjects who are past menarche
* Subjects give written or verbal assent, as applicable, and parents(s) or legal guardian(s) give written informed consent

Exclusion Criteria:

* Weight less than 15 kg
* History or presence of any condition that contraindicates routine dental care or use of local anesthetic
* Requires more than half cartridge of local anesthetic if weight is greater than or equal to 15 kg and less than 30 kg and more than one cartridge of local anesthetic if weight is greater than or equal to 30 kg, excluding supplemental injections
* Allergy or intolerance to lidocaine, epinephrine, sulfites, phentolamine, or topical benzocaine
* Has used any investigational drug and/or participated in any clinical study within 30 days of study drug administration
* Has participated in this study or any previous study of phentolamine mesylate for reversal of local soft tissue anesthesia (STA)
* Use of opioid-like analgesics within 24 hours prior to administration of local anesthetic
* Requires the use of local anesthetic other than lidocaine/epinephrine to perform the scheduled dental procedure
* Requires the use of nitrous oxide or sedatives to perform the scheduled dental procedure
* Any condition which, in the opinion of the Investigator, increases the risk to the subject of participating in the study or decreases the likelihood of compliance with the protocol

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2006-03; Study Completion 2006-08

PRIMARY OUTCOMES:
(All subjects) to evaluate the safety and tolerability of NV-101 as measured by: incidence, severity of adverse events
incidence, severity and duration of intraoral pain as measured by Wong Baker Pain Rating Scale
clinically significant changes in vital signs
clinically significant changes in oral cavity assessments
analgesics required for intraoral pain

SECONDARY OUTCOMES:
(For subjects 6 to 11 years of age who are trainable in standardized palpation procedure): to determine if NV-101 accelerates the time to normal tongue sensation as measured by standardized palpation procedure
for mandibular procedures, to determine if NV-101 accelerates the time to normal tongue sensation as measured by standardized palpation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mary Tavares, DDS, Principal Investigator — The Forsyth Institute
Locations (1):
- The Forsyth Institute, Boston, Massachusetts, United States